CLINICAL TRIAL: NCT02326493
Title: Tailor-CRT: Better Application of Cardiac Resynchronization Therapy by Automated and Improved Selection of Location and Timing of Stimulation
Brief Title: Tailor-CRT: Better Application of Cardiac Resynchronization Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 13-2-046
Record Dates: First submitted 2014-11-27; First posted 2014-12-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-09

CONDITIONS: Heart Failure; Left Bundle-Branch Block
Keywords: Cardiac Resynchronization Therapy; LV lead position; Device programming; Optimization; Vectorcardiography
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRT implantation (Experimental): Patients who have a class I indication for cardiac resynchronization therapy according to current international guidelines
  Interventions: Device: Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — A CRT device will be implanted while performing extra hemodynamic (LV dP/dtmax) and electrical (LVLED, VCG, and D-VCG) measurements. Devices and leads from various vendors will be used.

SUMMARY:
Approximately one third of patients treated with cardiac resynchronization therapy (CRT) do not derive any clinical benefit. CRT response can be improved by tailoring LV lead placement and programming of atrio-ventricular (AV) and inter-ventricular (VV) stimulation intervals to the individual patient. However, the best strategy to optimize lead positioning and device programming still remains to be established. Earlier work in our research group suggests that the vector cardiogram (VCG) can be used to determine the optimal LV lead position and AV- and VV-intervals, and pilot studies showed the feasibility to derive a VCG-like signal (D-VCG) from the implanted pacing electrodes. Other studies have suggested that the best position for the LV electrode is the region of latest electrical activation. The region of latest electrical activation can be identified by measuring the electrical delay on the LV lead (LVLED) during implantation. The objective of this study is to investigate whether D-VCG can be used to determine the optimal AV- and VV-interval and whether VCG and LVLED can be used to determine the optimal LV lead position.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is an established treatment for heart failure (HF) patients with severe left ventricular (LV) systolic impairment and delayed electrical impulse conduction through the ventricles, such as left bundle-branch block (LBBB). Since initial approval of the therapy over 10 years ago, there have been hundreds of thousands of implants worldwide. In The Netherlands, currently more than 2000 CRT devices are implanted each year. In a heart with LBBB, electrical activation of the lateral LV free wall is delayed, which leads to dyssynchronous and inefficient LV mechanical contraction and compromised LV pump function. The positive impact of CRT on LV pump function is attributed to paced pre-excitation of the delayed activated lateral LV wall. CRT is most commonly applied by pacing the right ventricle (RV) and LV lateral wall (almost) simultaneously. This corrects the abnormal LV electrical activation and resynchronizes LV mechanical contraction, which in turn results in improved LV pump function.

Despite the striking effectiveness of CRT, 30-50% of apparently suitable patients show little or no improvement. Previous studies have shown that the response to CRT can be improved by tailoring LV lead placement and programming of atrioventricular (AV) and inter-ventricular (VV) stimulation intervals to the individual patient. In clinical practice, echocardiographic techniques are the most widely employed for CRT optimization. However these techniques are subject to large measurement errors and inter- and intra-observer variability. A more accurate technique is invasive assessment of acute hemodynamic response to CRT, with the most widely used invasive hemodynamic parameter being the maximum rate of LV systolic pressure rise (LVdP/dtmax). However, the invasive and time-consuming nature of this approach limits its use in clinical practice. Thus, the best strategy to optimize lead positioning and device programming still remains to be established.

Earlier work in our research group suggests that the vectorcardiogram (VCG) can be used to determine the optimal LV lead position and AV- and VV-intervals, and pilot studies showed the feasibility to derive a VCG-like signal (D-VCG) from the implanted pacing electrodes. Other studies have suggested that the best position for the LV electrode is the region of latest electrical activation. The region of latest electrical activation can be identified by measuring the electrical delay on the LV lead (LVLED) during implantation. Validation of these techniques for tailoring LV lead positioning and AV- and VV- stimulation intervals to the individual patient, will provide non-invasive and easy methods to optimize CRT application and improve response rate.

The objective of this study is to investigate whether D-VCG can be used to determine the optimal AV- and VV-interval and whether VCG and LVLED can be used to determine the optimal LV lead position. Validation of these techniques for tailoring LV lead positioning and AV- and VV- stimulation intervals to the individual patient, will provide non-invasive and easy methods to optimize CRT application and improve response rate.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with NYHA functional class II-IV
* Left ventricular ejection fraction (LVEF) < 35%
* Left bundle-branch block (LBBB) with QRS duration > 120 ms
* In sinus rhythm

Exclusion Criteria:

* Atrial fibrillation
* ≥4 premature ventricular complexes on standard 12-lead ECG
* Age <18 years or > 80 years
* Incapable of giving informed consent
* Moderate to severe aortic valve stenosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Correlation between the increase in LV dP/dtmax and the D-VCG derived QRS area, obtained at different AV- and VV-intervals. | Acute measurements are performed for the duration of the CRT implantation procedure, an expected average of three hours
  The optimal AV- and VV-interval produces the maximal increase in LV dP/dtmax. It is investigated whether the maximal increase in LV dP/dtmax also corresponds to the minimal QRS area derived from the D-VCG. The correlations will be expressed by the Pearson Correlation coefficient.
Correlation between the increase in LV dP/dtmax and the LVLED or VCG derived QRS area, obtained at different potential LV lead positions | Acute measurements are performed for the duration of the CRT implantation procedure, an expected average of three hours
  The optimal LV lead position produces the maximal increase in LV dP/dtmax. It is investigated whether the maximal increase in LV dP/dtmax also corresponds to the longest LVLED or the minimal QRS area derived from the VCG. The correlations will be expressed by the Pearson Correlation coefficient.

SECONDARY OUTCOMES:
Correlations between QRS vector area, -angle and -amplitude derived from VCG and from D-VCG. | Acute measurements are performed for the duration of the CRT implantation procedure, an expected average of three hours
  The correlations will be expressed by the Pearson Correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Vernooy, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701
- [Background] European Heart Rhythm Association; European Society of Cardiology; Heart Rhythm Society; Heart Failure Society of America; American Society of Echocardiography; American Heart Association; European Association of Echocardiography; Heart Failure Association; Daubert JC, Saxon L, Adamson PB, Auricchio A, Berger RD, Beshai JF, Breithard O, Brignole M, Cleland J, Delurgio DB, Dickstein K, Exner DV, Gold M, Grimm RA, Hayes DL, Israel C, Leclercq C, Linde C, Lindenfeld J, Merkely B, Mont L, Murgatroyd F, Prinzen F, Saba SF, Shinbane JS, Singh J, Tang AS, Vardas PE, Wilkoff BL, Zamorano JL. 2012 EHRA/HRS expert consensus statement on cardiac resynchronization therapy in heart failure: implant and follow-up recommendations and management. Heart Rhythm. 2012 Sep;9(9):1524-76. doi: 10.1016/j.hrthm.2012.07.025. No abstract available. PMID 22939223
- [Background] Auricchio A, Prinzen FW. Non-responders to cardiac resynchronization therapy: the magnitude of the problem and the issues. Circ J. 2011;75(3):521-7. doi: 10.1253/circj.cj-10-1268. Epub 2011 Feb 11. PMID 21325727
- [Background] Cazeau S, Leclercq C, Lavergne T, Walker S, Varma C, Linde C, Garrigue S, Kappenberger L, Haywood GA, Santini M, Bailleul C, Daubert JC; Multisite Stimulation in Cardiomyopathies (MUSTIC) Study Investigators. Effects of multisite biventricular pacing in patients with heart failure and intraventricular conduction delay. N Engl J Med. 2001 Mar 22;344(12):873-80. doi: 10.1056/NEJM200103223441202. PMID 11259720
- [Background] Auricchio A, Stellbrink C, Block M, Sack S, Vogt J, Bakker P, Klein H, Kramer A, Ding J, Salo R, Tockman B, Pochet T, Spinelli J. Effect of pacing chamber and atrioventricular delay on acute systolic function of paced patients with congestive heart failure. The Pacing Therapies for Congestive Heart Failure Study Group. The Guidant Congestive Heart Failure Research Group. Circulation. 1999 Jun 15;99(23):2993-3001. doi: 10.1161/01.cir.99.23.2993. PMID 10368116
- [Background] Auricchio A, Ding J, Spinelli JC, Kramer AP, Salo RW, Hoersch W, KenKnight BH, Klein HU. Cardiac resynchronization therapy restores optimal atrioventricular mechanical timing in heart failure patients with ventricular conduction delay. J Am Coll Cardiol. 2002 Apr 3;39(7):1163-9. doi: 10.1016/s0735-1097(02)01727-8. PMID 11923041
- [Background] Butter C, Auricchio A, Stellbrink C, Fleck E, Ding J, Yu Y, Huvelle E, Spinelli J; Pacing Therapy for Chronic Heart Failure II Study Group. Effect of resynchronization therapy stimulation site on the systolic function of heart failure patients. Circulation. 2001 Dec 18;104(25):3026-9. doi: 10.1161/hc5001.102229. PMID 11748094
- [Background] Sawhney NS, Waggoner AD, Garhwal S, Chawla MK, Osborn J, Faddis MN. Randomized prospective trial of atrioventricular delay programming for cardiac resynchronization therapy. Heart Rhythm. 2004 Nov;1(5):562-7. doi: 10.1016/j.hrthm.2004.07.006. PMID 15851220
- [Background] Morales MA, Startari U, Panchetti L, Rossi A, Piacenti M. Atrioventricular delay optimization by doppler-derived left ventricular dP/dt improves 6-month outcome of resynchronized patients. Pacing Clin Electrophysiol. 2006 Jun;29(6):564-8. doi: 10.1111/j.1540-8159.2006.00402.x. PMID 16784420
- [Background] Hardt SE, Yazdi SH, Bauer A, Filusch A, Korosoglou G, Hansen A, Bekeredjian R, Ehlermann P, Remppis A, Katus HA, Kuecherer HF. Immediate and chronic effects of AV-delay optimization in patients with cardiac resynchronization therapy. Int J Cardiol. 2007 Feb 14;115(3):318-25. doi: 10.1016/j.ijcard.2006.03.015. Epub 2006 Aug 7. PMID 16891011
- [Background] Delnoy PP, Ottervanger JP, Luttikhuis HO, Vos DH, Elvan A, Ramdat Misier AR, Beukema WP, Steendijk P, van Hemel NM. Pressure-volume loop analysis during implantation of biventricular pacemaker/cardiac resynchronization therapy device to optimize right and left ventricular pacing sites. Eur Heart J. 2009 Apr;30(7):797-804. doi: 10.1093/eurheartj/ehp011. Epub 2009 Feb 7. PMID 19202156
- [Background] Derval N, Steendijk P, Gula LJ, Deplagne A, Laborderie J, Sacher F, Knecht S, Wright M, Nault I, Ploux S, Ritter P, Bordachar P, Lafitte S, Reant P, Klein GJ, Narayan SM, Garrigue S, Hocini M, Haissaguerre M, Clementy J, Jais P. Optimizing hemodynamics in heart failure patients by systematic screening of left ventricular pacing sites: the lateral left ventricular wall and the coronary sinus are rarely the best sites. J Am Coll Cardiol. 2010 Feb 9;55(6):566-75. doi: 10.1016/j.jacc.2009.08.045. Epub 2009 Nov 20. PMID 19931364
- [Background] van Campen CM, Visser FC, de Cock CC, Vos HS, Kamp O, Visser CA. Comparison of the haemodynamics of different pacing sites in patients undergoing resynchronisation treatment: need for individualisation of lead localisation. Heart. 2006 Dec;92(12):1795-800. doi: 10.1136/hrt.2004.050435. Epub 2006 Jun 27. PMID 16803940
- [Background] Cuoco FA, Gold MR. Optimization of cardiac resynchronization therapy: importance of programmed parameters. J Cardiovasc Electrophysiol. 2012 Jan;23(1):110-8. doi: 10.1111/j.1540-8167.2011.02235.x. Epub 2011 Dec 21. PMID 22188487
- [Background] van Deursen CJ, Strik M, Rademakers LM, van Hunnik A, Kuiper M, Wecke L, Crijns HJ, Vernooy K, Prinzen FW. Vectorcardiography as a tool for easy optimization of cardiac resynchronization therapy in canine left bundle branch block hearts. Circ Arrhythm Electrophysiol. 2012 Jun 1;5(3):544-52. doi: 10.1161/CIRCEP.111.966358. Epub 2012 Apr 24. PMID 22534251
- [Background] Gold MR, Birgersdotter-Green U, Singh JP, Ellenbogen KA, Yu Y, Meyer TE, Seth M, Tchou PJ. The relationship between ventricular electrical delay and left ventricular remodelling with cardiac resynchronization therapy. Eur Heart J. 2011 Oct;32(20):2516-24. doi: 10.1093/eurheartj/ehr329. Epub 2011 Aug 29. PMID 21875862
- [Background] Kandala J, Upadhyay GA, Altman RK, Parks KA, Orencole M, Mela T, Kevin Heist E, Singh JP. QRS morphology, left ventricular lead location, and clinical outcome in patients receiving cardiac resynchronization therapy. Eur Heart J. 2013 Aug;34(29):2252-62. doi: 10.1093/eurheartj/eht123. Epub 2013 Apr 9. PMID 23571836